CLINICAL TRIAL: NCT03391999
Title: (Danish): Sundhed, Trivsel og Læring på HHX og HTX, Erhvervsskolerne i Aars
Brief Title: Health-Related Quality of Life in Upper Secondary Schools in Denmark
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Karin Dam Petersen, Associate Professor, Aalborg University
Other Study IDs: AalborgU
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2019-07

CONDITIONS: Quality of Life
Keywords: Mental Health, Physical Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A questionnaire; CHU9D — Measuring Health Related Quality of Life

SUMMARY:
Measuring Quality of Life in an upper secondary school in Denmark

DETAILED DESCRIPTION:
The Child Health Utility 9 Dimension (CHU9D) is a relatively new health-related quality of life (HRQoL) instrument for use in children and young people. CHU9D has recently been translated and linguistic validated into Danish.

The objective of this study is twofold. Firstly, the investigators wants to examine the feasibility of using the Danish version of CHU9D to assess the HRQoL in young adults. Secondly, the investigators wants to analyse the association of wellbeing, happiness with the school and the learning environment with the students HRQoL in the Northern Danish Region of Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Students at the Higher Commercial Examination (HHX) and Higher Technical Examination (HTX) at the Technical College in Aars.

Exclusion Criteria:

* There will be no exclusion criteria concerning diseases or conditions for these school students.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young adults enrolled at the Technical College in Aars
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-10-15 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
QALY | 3-5 years
  Quality Adjusted Life Years

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Gregersen, PhD, Study Director — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Only sharing IPD with the upper secondary school and my research group

REFERENCES:
- [Derived] Petersen KD, Ratcliffe J, Chen G, Serles D, Frosig CS, Olesen AV. The construct validity of the Child Health Utility 9D-DK instrument. Health Qual Life Outcomes. 2019 Dec 23;17(1):187. doi: 10.1186/s12955-019-1256-0. PMID 31870369